CLINICAL TRIAL: NCT06208072
Title: The Predictive Role of Urinary Proteomics in Blood Pressure Response of Obese Hypertensive Treated With Irbesartan or Eplerenone.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor Of Cardiology, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PREDICT-HTN
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Primary Hypertension; Obesity
Keywords: Hypertension; Obesity; Urinary Proteomics; Proteomic Analysis; Biomarkers
MeSH Terms: conditions — Essential Hypertension; Obesity; Hypertension | interventions — Irbesartan; Eplerenone

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomized into two arms. One arm will receive treatment with Irbesartan 150mg once daily and the second arm will receive treatment with Eplerenone 25mg twice daily. Blood pressure response will be assessed after 8 weeks. For both arms peptide differences will be assessed through proteomic analysis in responders and non responders in each individual arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irbesartan group (Active Comparator): Randomized obese hypertensive patients will receive treatment with oral Irbesartan 150mg once daily for 8 weeks. Blood pressure response will be assessed at that time.
  Interventions: Drug: Irbesartan 150mg
- Eplerenone group (Active Comparator): Randomized obese hypertensive patients will receive treatment with oral Eplerenone twice daily for 8 weeks. Blood pressure response will be assessed at that time.
  Interventions: Drug: Eplerenone 25 mg

INTERVENTIONS:
Drug: Irbesartan 150mg — Irbesartan group will be treated with Irbesartan 150mg once daily for a total of 8 weeks.
  Other Names: I
  Arms: Irbesartan group
Drug: Eplerenone 25 mg — Eplerenone group will be treated with Eplerenone 25mg twice daily for a total of 8 weeks
  Other Names: E
  Arms: Eplerenone group

SUMMARY:
Despite the available means of treating primary arterial hypertension, the prevalence of hypertensive patients with inadequately controlled blood pressure levels, remains high. The identification of biomarkers with prognostic and predictive roles seems to play an important role in the management of hypertensive patients. Proteomic analysis studies provide encouraging results in the identification of such biomarkers.

The goal of this clinical study is to is to highlight peptides through urinary proteomic analysis of obese hypertensive patients, capable of predicting blood pressure response, following treatment with irbesartan or eplerenone.

DETAILED DESCRIPTION:
Background :

Hypertension remains the most prevalent modifiable risk factor associated with cardiovascular morbidity and mortality, however un-optimally treated hypertension prevalence remains alarmingly high. Variable blood pressure response to pharmacological treatment, physician inertia and lack of patient's compliance due to polypharmacy, are the main reasons behind non optimal blood pressure treatment. The multifactorial nature of hypertension has long been described, with various environmental, genetic and epi-genetic factors involved in its pathogenesis and progression. Therefore, scientific interest is starting to shift towards precision medicine, as a medical model for disease prevention and tailored treatment that incorporates individual, genetic, environmental and experiential variability. Το this end, proteomic analysis is an emerging representative in the research of predictive biomarkers.

Proteomic analysis consists of the qualitive and quantitative analysis of the final proteins in bodily fluids. A simplified approach constitutes of sample acquisition, protein extraction and separation through high-resolution electrophoresis and chromatography-based techniques, protein sequence determination with mass spectrometry-based analysis and protein identification with bioinformatic techniques in referential databases. Various small scale clinical trials have highlighted the clinical significance if proteomic analysis, ranging from identifying biomarkers able to determine the blood pressure response following treatment with spironolactone in patients with resistant hypertension, predicting pre-eclampsia through the urinary proteome even in early stages of gestation.

Obesity and essential hypertension are two pathological entities that often coexist. Data from the Framingham study suggesting a twofold risk of obese patients developing hypertension compared to underweight ones, while similar associations have been described by the NHANES III, MONICA, and Health, Aging and Body Composition Study studies, between increases in blood pressure, as a result of increases in BMI, waist circumference, and visceral fat, respectively. The mechanisms through which obesity leads to the development of hypertension, are a complex pathophysiological phenomenon under constant research and study, including the activation of the Sympathetic Nervous System, disorder of renal sodium excretion, excessive renin-angiotensin-aldosterone axis activation and endothelial dysfunction. Angiotensin 2 receptor blockers like Irbesartan, have long been used as first-line pharmacological treatment, however clinical trials including ASPIRANT, PATHWAY-2, and RALES study, have highlighted the role of aldosterone receptor blockers in obese hypertensive patients. Spironolactone and eplerenone are the main oral representatives of this group, with the latter showing less frequent side effects as well as higher binding specificity for the mineralocorticoid- receptor.

Aim of the study:

The main purpose of this study is to investigate the potential predictive role of urinary proteomics, in blood pressure response of obese hypertensive patients, after treatment with irbesartan or eplerenone. This hypothesis may lead to the emergence of urinary biomarkers able to predict blood pressure response in obese hypertensive patients.

Study design:

In this interventional study, untreated obese hypertensive patients will be randomized to two pharmacological treatment arms. Blood pressure response will be assessed based on a baseline visit prior to the initiation of pharmacological treatment and a follow-up visit after an 8-week interval. Patients will be categorized as either responders or non-responders based on the changes in their blood pressure levels. The analysis of patients' baseline urinary samples will be conducted using Liquid Chromatography with tandem mass spectrometry (LC-MS/MS). The examination of individual urinary peptides, along with the evaluation of blood pressure response, will be employed to pinpoint distinct urinary proteins that can act as indicators predicting the response to blood pressure alterations after pharmacological treatment.

Methods:

A total of 50 untreated obese hypertensive adults, will be randomized to irbesartan 150mg once daily, or eplerenone 25mg twice daily.

Patients will undergo a detailed medical history questionnaire and clinical-laboratory examination, in order to ensure that the inclusion and exclusion criteria are met. For inclusion in the study, signed informed consent will be required, after detailed briefing on the study procedure and objectives, as well as potential risks. Ethics approval has been obtained from the hospital's ethical committee board.

Baseline blood pressure levels will be determined with ambulatory blood pressure measurement (ABPM), office blood pressure measurement (OBP) and home blood pressure measurement (HBP). Before treatment initiation, a urinary sample will be collected and stored under appropriate conditions, until subjected to proteomic analysis. Patient data will be recorded anonymously in an electronic database, through which randomization of patients will be carried out. Following randomization, medication stored appropriately on-site, will be administered to each patient.

The participants will undergo a follow-up visit after 8 weeks, where blood pressure response will be determined with ABPM, OBP and HBP. Adherence to treatment will be determined though a medication diary, provided at baseline visit. Patients with ≥ 5mmHg reduction in systolic mean ABPM and/or ≥10mmHg systolic OBP reduction will be considered responders to the corresponding treatment.

Stored urinary samples will undergo liquid chromatography with tandem mass spectrometry (LC-MS/MS) analysis. Data will be processed and cross-referenced with bioinformatics software and databases for protein identification. To establish the certainty of the protein identification false discovery rate (FDR) validation will be based on q value, with target FDR: 0.05. Peptide distribution of intensity between responders and non responders will be assessed, to establish differential expression in each arm. Differential expression will be measured in fold change, as the relative difference in protein abundance between the two conditions. Student's t-test or Mann Whitney non-parametric test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Systolic office blood pressure 140-179mmHg and/or diastolic office blood pressure 90-119mmHg
* Mean systolic 24h ABPM >130mmHg and/or mean diastolic ABPM >80mmHg
* Obese patient with BMI 30-39.99kg/m2
* Signed informed consent

Exclusion Criteria:

* Participation in an Investigational Medicinal Product (IMP) or invasive device clinical trial during the study or in the last 6 months
* Patient with secondary arterial hypertension
* Patient with a history within 6 months of: Myocardial infarction, Unstable angina, Stroke
* Patient with type 1 diabetes
* Patient with systolic heart failure EF≤40%
* Patient with chronic kidney disease (eGFR<45mL/min/1.73m2)
* Patient with bilateral renal artery stenosis
* Patient with hyperkalemia (>5.5 mEq/L)
* Patient with hemodynamically significant valvular heart disease
* Patient with Addison's disease
* Female patient in pregnancy or caesarean section or female patient planning pregnancy.
* Planned surgery or cardiovascular surgery in the next 6 months
* Patient with absolute contraindication to any EDPS
* Patient who needs to receive study medication for a different reason
* Patient with neoplasia undergoing treatment (radiotherapy, chemotherapy, immunotherapy)
* Patient with synchronous systemic disease with a survival expectancy less than the end of the study
* Any condition that, in the judgment of the investigator, may adversely affect the efficacy and/or safety of the Investigational Medicinal Products (IEDs) (alcohol abuse, drug use, mental retardation)
* Patient who has received treatment with systemic corticosteroids at least 3 months before joining the study
* Patient receiving α-blockers with the exception of alfuzosin and tamsulosin for prostatic symptoms

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Urinary peptide differential expression between responders and non-responders, in patients treated with Irbesartan | 8 weeks
  Utilizing liquid chromatography with tandem mass spectrometry (LC/MS-MS) the relative difference in protein abundance between responders and non-responders will be measured, expressed in fold change. Peptides with statistically significant differential expression between the two groups, may be used as urinary biomarkers for blood pressure response.
Urinary peptide differential expression between responders and non-responders, in patients treated with Eplerenone | 8 weeks
  Utilizing LC/MS-MS, the relative difference in protein abundance between responders and non-responders will be measured, expressed in fold change. Peptides with statistically significant differential expression between the two groups, may be used as urinary biomarkers for blood pressure response.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Tsioufis, Prof, Principal Investigator — First University Cardiology Clinic, Hippocration General Hospital of Athens
Locations (1):
- Hypertension Unit, A' University Cardiology Clinic, Hippocration General Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitt J, Fox R, Tucker KL, McManus RJ. New Approaches in Hypertension Management: a Review of Current and Developing Technologies and Their Potential Impact on Hypertension Care. Curr Hypertens Rep. 2019 Apr 25;21(6):44. doi: 10.1007/s11906-019-0949-4. PMID 31025117
- [Background] Mills KT, Stefanescu A, He J. The global epidemiology of hypertension. Nat Rev Nephrol. 2020 Apr;16(4):223-237. doi: 10.1038/s41581-019-0244-2. Epub 2020 Feb 5. PMID 32024986
- [Background] Manolis AJ, Poulimenos LE, Kallistratos MS, Gavras I, Gavras H. Sympathetic overactivity in hypertension and cardiovascular disease. Curr Vasc Pharmacol. 2014 Jan;12(1):4-15. doi: 10.2174/15701611113119990140. PMID 23905597
- [Background] Tsioufis C, Kordalis A, Flessas D, Anastasopoulos I, Tsiachris D, Papademetriou V, Stefanadis C. Pathophysiology of resistant hypertension: the role of sympathetic nervous system. Int J Hypertens. 2011 Jan 20;2011:642416. doi: 10.4061/2011/642416. PMID 21331155
- [Background] Navajas R, Corrales F, Paradela A. Quantitative proteomics-based analyses performed on pre-eclampsia samples in the 2004-2020 period: a systematic review. Clin Proteomics. 2021 Jan 26;18(1):6. doi: 10.1186/s12014-021-09313-1. PMID 33499801
- [Background] Martin-Lorenzo M, Martinez PJ, Baldan-Martin M, Lopez JA, Minguez P, Santiago-Hernandez A, Vazquez J, Segura J, Ruiz-Hurtado G, Vivanco F, Barderas MG, Ruilope LM, Alvarez-Llamas G. Urine Haptoglobin and Haptoglobin-Related Protein Predict Response to Spironolactone in Patients With Resistant Hypertension. Hypertension. 2019 Apr;73(4):794-802. doi: 10.1161/HYPERTENSIONAHA.118.12242. PMID 30712426
- [Background] Correa Rojo A, Heylen D, Aerts J, Thas O, Hooyberghs J, Ertaylan G, Valkenborg D. Towards Building a Quantitative Proteomics Toolbox in Precision Medicine: A Mini-Review. Front Physiol. 2021 Aug 26;12:723510. doi: 10.3389/fphys.2021.723510. eCollection 2021. PMID 34512391
- [Background] Alharbi RA. Proteomics approach and techniques in identification of reliable biomarkers for diseases. Saudi J Biol Sci. 2020 Mar;27(3):968-974. doi: 10.1016/j.sjbs.2020.01.020. Epub 2020 Jan 27. PMID 32127776
- [Background] Schessner JP, Voytik E, Bludau I. A practical guide to interpreting and generating bottom-up proteomics data visualizations. Proteomics. 2022 Apr;22(8):e2100103. doi: 10.1002/pmic.202100103. Epub 2022 Feb 15. PMID 35107884